CLINICAL TRIAL: NCT06520098
Title: Benefit of Venetoclax Addition ("Benefit VA") in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: A Randomized Phase II Study Of Bruton Tyrosine Kinase Inhibitor With Or Without Venetoclax In Veterans With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Acronym: Benefit VA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEMA-001-23S
Record Dates: First submitted 2024-02-12; First posted 2024-07-25 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma | interventions — venetoclax; ibrutinib; acalabrutinib; zanubrutinib

STUDY DESIGN:
Intervention Model Description: The addition of Venetoclax to BTKi for 12 months in anticipated to improve both the clinical response rates and the quality of life of patients as compared to indefinite use of BTKi monotherapy in CLL/SLL patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A : Continue BTKi single agent (Active Comparator): Continue BTKi single agent (monotherapy) Standard Intervention
  Interventions: Drug: Ibrutinib, Acalabrutinib, Zanubrutinib
- Arm B : BTKi + Venetoclax for 12 cycles, then discontinue (Experimental): BTKi + Venetoclax for 12 cycles, then discontinue Experimental Intervention
  Interventions: Drug: Venetoclax; Drug: Ibrutinib, Acalabrutinib, Zanubrutinib

INTERVENTIONS:
Drug: Venetoclax — VENCLEXTA is indicated for the treatment of patients with chronic lymphocytic leukemia (CLL) with 17p deletion, as detected by an FDA approved test, who have received at least one prior therapy.
  Other Names: VENCLEXTA
  Arms: Arm B : BTKi + Venetoclax for 12 cycles, then discontinue
Drug: Ibrutinib, Acalabrutinib, Zanubrutinib — IMBRUVICA is a kinase inhibitor Acalabrutinib is a selective, irreversible small molecule inhibitor of BTK. Zanubrutinib is BTK inhibitors
  Other Names: IMBRUVICA, CALQUENCE, BRUKINSA

SUMMARY:
People who have chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) are often treated with ibrutinib, acalabrutinib, or zanubrutinib. These are pills that are taken by mouth. This type of pill is called "Bruton Tyrosine Kinase Inhibitor" or BTKi. Another treatment for CLL/SLL is a different pill called venetoclax.

The purpose of this study is to compare continuing the current treatment with BTKi alone, as long as it is working, to another arm of treatment which adds venetoclax to the current treatment (BTKi), for one year. After one year, both pills in this arm of treatment would be stopped and the participants will be closely monitored.

DETAILED DESCRIPTION:
People who have chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) are often treated with ibrutinib, acalabrutinib, or zanubrutinib. These are pills that are taken by mouth. This type of pill is called a "Bruton Tyrosine Kinase Inhibitor" or BTKi. Another treatment for CLL/SLL is a different pill called venetoclax.

People with CLL/SLL who are currently taking BTKi as their treatment must continue to take the medicine for the rest of their lives (unless it is no longer working or causing difficult side effects).

New studies tested the combination of BTKi and venetoclax for one to two years, and showed that it was a very effective treatment, and allowed patients to stop therapy.

The investigators don't know if adding venetoclax in patients who have already taken BTKi therapy for at least six months and who are responding to it will help control the CLL/SLL better and if it will allow them to stop treatment safely. Also, the investigators don't know how the side effects and effectiveness of the combination will be in Veterans. The investigators also don't know how a patient's quality of life will be affected if they continue BTKi by itself or if they take the combination and then are able to stop treatment.

If participants meet the eligibility criteria, they will be randomly assigned a study treatment. This study has 2 main study groups:

ARM A (BTKI ALONE): There will be about 50 people in this group.

ARM B (BTKI PLUS VENETOCLAX): There will be about 50 people in this group.

The participants will not be charged for any treatments or procedures that are part of this study. If participants usually pay co-payments for VA care and medications, they will still pay these co-payments for VA care and medications that are not part of this study.

ELIGIBILITY:
Inclusion Criteria:

* CLL or SLL diagnosis
* Patients must have been diagnosed with CLL (> 5000 B-cells per uL of peripheral blood at any point during the course of their disease) or small lymphocytic lymphoma (SLL) with <5000 B-cells per µL of blood but with disease-associated lymphadenopathy by 2018 IWCLL criteria.
* Prior treatment
* Patients must be currently receiving CLL/SLL directed therapy with a BTKi (i.e., ibrutinib, acalabrutinib, zanubrutinib) for at least six months.
* The dose of BTKi must be stable for at least the past three months.
* Age 18 years
* ECOG performance status 0-2
* Detectable or measurable CLL/SLL in blood or imaging during the screening period.

Detectable CLL/SLL in the blood is defined either by elevation in absolute lymphocyte count or by diagnostic flow cytometry from blood demonstrating presence of CLL cells.

* Low TLS risk, defined as having all lymph nodes less than 5 cm in diameter (radiographically) and absolute lymphocyte count less than 25 x 109/L in blood, within 30 days of enrollment.
* Required initial laboratory values
* Absolute Neutrophil Count (ANC) 1,000/mm3 except if due to bone marrow involvement
* Platelet Count (untransfused) 30,000/mm3 except if due to bone marrow involvement
* Calc. Creatinine Clearance 40 mL/min (by Cockcroft-Gault)
* Bilirubin 1.5 x upper limit of normal (ULN) except if due to liver involvement, hemolysis, or Gilbert's disease
* AST / ALT 2.5 x upper limit of normal (ULN) except if due to liver involvement
* Other
* Patients must be able to swallow oral medications and not have the following conditions: disease significantly affecting gastrointestinal absorption, resection of the stomach or small bowel, partial or complete bowel obstruction.
* Patients must be able to receive either a xanthine oxidase inhibitor or rasburicase

Exclusion Criteria:

* Prior treatment
* Patients must not have progression of CLL/SLL on BTKi therapy prior to initiation of the study therapy.
* Patients must not have received the combination of BTKi + venetoclax previously.
* Comorbid conditions or other active diseases
* Patients must not have any history of Richter's transformation or prolymphocytic leukemia.
* If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable and be on suppressive therapy, if indicated.
* Please note: IVIG can cause a false positive hepatitis B serology. If patients receiving routine IVIG have core antibody or surface antigen positivity without evidence of active viremia (negative hepatitis B DNA) they may still participate in the study, must have hepatitis serologies and hepatitis B DNA monitored periodically by the treating physician.
* If history of hepatitis C virus (HCV) infection, must be treated with undetectable HCV viral load.
* Patients with Class III or Class IV heart failure by New York Heart Association, those with unstable angina, and those with uncontrolled arrhythmia are not eligible.
* Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy are eligible for this trial.
* Concomitant medications
* Patients must not be receiving active systemic anticoagulation with heparin or warfarin. Patients on warfarin must discontinue the drug for at least 10 days prior to registration on the study.
* Chronic concomitant treatment with strong inhibitors of CYP3A4/5 is not recommended on this study. Patients on strong CYP3A inhibitors must discontinue the drug for 14 days prior to registration on the study or discuss with the study principal investigator.
* Chronic concomitant treatment with strong CYP3A4/5 inducers is not recommended. Patients must discontinue the drug 14 days prior to registration on the study or discuss with the study principal investigator.
* Patients must not require more than 20 mg prednisone or equivalent corticosteroid daily.
* Patients must not have uncontrolled active systemic infection requiring intravenous antibiotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate complete response (CR) rate, per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria, 2018 | 24-36 months
  The addition of Venetoclax to BTKi for 12 months will improve CR compared to use of BTKi alone in CLL/SLL patients who are already receiving BTKi therapy as treatment.

SECONDARY OUTCOMES:
CLL/SLL patients' experience through patient reported outcome (PRO) measures of fatigue (a key secondary objective) | 24-36 months
  The addition of Venetoclax to BTKi for 12 months is anticipated to improve cancer-related fatigue as compared to use of BTKi alone in CLL/SLL patients. FACIT-Fatigue PRO instrument will be used.
Undetectable minimal residual disease (MRD) in the peripheral blood (PB). | 24-36 months
  Use residual disease (MRD) assays in the peripheral blood (PB).
Safety and adverse events, measured by Common Terminology Criteria for Adverse Events (CTCAE). | 24-36 months
  Safety and adverse events, measured by Common Terminology Criteria for Adverse Events (CTCAE).
Overall response rate (ORR), per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria, 2018. | 24 - 36 months
  Overall response rate (ORR), per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria, 2018.
Measure financial toxicity (FT) in CLL/SLL patients | 24-36 months
  The addition of Venetoclax to BTKi for 12 months is anticipated to improve cancer-related fatigue as compared to use of BTKi alone in CLL/SLL patients. FACT-COST PRO instrument will be used. The score ranges between 0 and 44, and a higher score implies better financial well-being.
CLL/SLL patients' experience through patient reported outcome (PRO) QoL | 24-36 months
  The addition of Venetoclax to BTKi for 12 months is anticipated to improve of cancer-related fatigue as compared to use of BTKi alone in CLL/SLL patients. Aggregate scores from PRO instruments (QLQ-C30, QLQ-CLL17) will be used. These multi-item scales range in score from 0 to 100. A high score on these scales represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Kambhampati, MD MBBS, Principal Investigator — Kansas City VA Medical Center, Kansas City, MO
Locations (4):
- United States (4):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No